CLINICAL TRIAL: NCT05546528
Title: Photobiomodulation Efficacy of Major Salivary Glands in Children With Caries Activity: Study Protocol for Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Trial
Brief Title: Photobiomodulation on Major Salivary Glands in Children With Caries Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMBSalivaCaries
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Caries,Dental
Keywords: dental caries; photobiomodulation; salivary flow
MeSH Terms: conditions — Dental Caries | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: two groups: 1) the photobiomodulation experimental group (G1) , 2) the photobiomodulationn placebo group (G2) .
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the researcher responsible for applying the laser will know which treatment was assigned to each participant. The researcher responsible for data collection will be blinded to the type of treatment received. The participant will be blind. The treatment with the control group will simulate the laser in operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photobiomodulation (Experimental): photobiomodulation application with the Laser Therapy XT device
  Interventions: Device: Photobiomodulation
- photbiomodulation-sham (Sham Comparator): photobiomodulation application with the Laser Therapy XT device off
  Interventions: Device: Photobiomodulation- Sham

INTERVENTIONS:
Device: Photobiomodulation — G1 will receive the photobiomodulation application with the Laser Therapy XT device, (DMC, São Paulo, Brazil). The laser will be applied for 60 seconds per point, in 2 extraoral points and 2 intraoral points in the region of the parotid glands bilaterally, as well as 1 extraoral point for the submandibular and sublingual glands (totaling 16 points).
  Arms: photobiomodulation
Device: Photobiomodulation- Sham — G2 will receive the photobiomodulation application with the Laser Therapy XT device off. The laser off will be applied for 60 seconds per point, in 2 extraoral points and 2 intraoral points in the region of the parotid glands bilaterally, as well as 1 extraoral point for the submandibular and sublingual glands (totaling 16 points).
  Arms: photbiomodulation-sham

SUMMARY:
The purpose of this trial is to evaluate the efficacy of photobiomodulation of the major salivary glands on salivary parameters in children with caries activity.

DETAILED DESCRIPTION:
Dental caries represents one of the most prevalent diseases among children around the world. Saliva plays a preponderant role in the process of demineralization- remineralization of the dental surface. Patient salivary characteristics, such as flow rate, pH, and buffering capacity, provide relevant information about patient's risk for developing carious lesions. Photobiomodulation has shown promising results to improve salivary flow rate, as well as buffer capacity in the adult population. The purpose of this trial is to evaluate the efficacy of photobiomodulation of the major salivary glands on salivary parameters in children with caries activity.

Methods: This protocol details a randomized, double-blind, parallel-group, controlled trial evaluating salivary parameters through photobiomodulation in children. Seventy-eight 6- to 12-year-old participants will be randomly divided in two groups: 1) the photobiomodulation experimental group (G1) (n=39), 2) the photobiomodulationn placebo group (G2) (n=39). Infrared light will be applied in 16 intra and extraoral points and the placebo, respectively. The unstimulated salivary sample will be taken before and immediately after the application once a week, for three consecutive weeks. Salivary samples will be analyzed for flow rate, pH and buffering capacity. The primary outcomes are difference in salivary flow rates between the G1 and the G2. The secondary outcomes are difference in salivary pH and buffering capacity between the G1 and the G2 group.

ELIGIBILITY:
nclusion criteria

* Individuals of both sexes, between 6 and 12 years old with mixed dentition.
* Participants diagnosed with the presence of at least one active caries lesion
* Good general health, without systemic or local diseases that affect salivary secretions.

Exclusion criteria

* Participants with severe active cavitated lesions with pulpal symptoms.
* Plans of the family nucleus to move for the duration of the study.
* Patients with a diagnosis of hyposalivation or xerostomia
* Presence of fixed appliances.
* Physical disability that interferes with oral or intellectual hygiene to answer the questionnaire.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Salivary flow | three weeks
  Saliva flow rate will be estimated by asking the children to salivate into the plastic cylinders (previously weighed) for 5 minutes. Next, these plastic cylinders (containing the saliva) will be weighed and the flow rate in g/ml will be calculated, which is equivalent to ml/min,

SECONDARY OUTCOMES:
Saliva pH | three weeks
  aliva pH will be measured using a previously calibrated digital pH meter

CONTACTS AND LOCATIONS:
Locations (1):
- Magdalena San-Martín, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No